CLINICAL TRIAL: NCT04971174
Title: Short & Medium Term Outcomes of Periodontal Regenerative Procedures. A Two-part Study With a) Analysis of Periodontal Records of a Cohort of Periodontitis Patients and b) a Single Visit Recall and Comprehensive Periodontal Re-evaluation
Brief Title: Outcomes of Periodontal Regenerative Treatment
Status: Enrolling by invitation | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 280800
Record Dates: First submitted 2021-06-22; First posted 2021-07-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Periodontitis; Intrabony Periodontal Defect; Periodontal Regeneration
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this recall study is to evaluate outcomes of surgical regenerative treatment of periodontal defects in a cohort of patient previously treated for gum disease at the Royal London Hospital as part of their periodontal care.

DETAILED DESCRIPTION:
This study will be divided in two parts:

Part 1: a retrospective analysis of short-term outcomes of periodontal regenerative procedures undertaken at the Barts Royal London Dental Hospital (RLDH); Part 2: a single recall visit study in which patients identified through part 1 and willing to consent for the study will be reassessed for medium-term outcomes of the regenerative procedures previously undertaken.

For part 1 historic data will be collected from available dental records at RLDH and divided in:

* Timepoint 0: the latest available full mouth periodontal assessment before surgery and x-ray of site/s needing surgical intervention
* Timepoint 1: the latest available full mouth periodontal assessment after surgery and x-ray of same site/s at Timepoint 0

For part 2 data will be collected from patients identified through part 1 and willing to give consent for a single study recall visit:

•Timepoint 2: single study outcome recall visit (full mouth periodontal assessment and x-ray of same site/s at Timepoint 0).

Due to the nature of the study, the time elapsed between Timepoint 0 and Timepoint 2 can vary between 1 and 4 years.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for part 1 of the study:

* Patient age 18 and older
* Patients that received periodontal regenerative surgical treatment at Barts RLDH from January 2017 to January 2019 with and without the use of any biomaterials, bone graft/substitute and membrane or combinations of those.
* Available full periodontal examination records after non surgical therapy to serve as a baseline for the study and not beyond 12 months before surgery
* Available radiographic examination of the tooth treated with surgical regenerative procedure at initial examination or after non surgical therapy to serve as a baseline for the study.

Additional inclusion criteria for part 2:

-Patient able and willing to give informed consent

Exclusion Criteria:

Exclusion criteria for part 1:

* All the patients that do not match the inclusion criteria will be excluded from part 1.
* Patients that received regenerative surgical treatment for the management of gingival recession.

Exclusion criteria for part 2:

* Unable or unwilling to give consent
* Pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cohort of patients that underwent surgical periodontal regenerative treatment at RLDH between January 2017 and January 2019 will be the study population for part 1 of the study.
  For the part 2 of the study these patients will be contacted and asked to participate in the recall study. The patients willing to participate into the single recall visit outcome study will form the study population for part 2.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
% of patients with pocket closure at worst site per mouth for intrabony defects | Through study completion, an average of 2 years
  Pocket closure is defined as PPD < and = 4 mm with no bleeding on probing (BoP)

SECONDARY OUTCOMES:
% of patients with pocket closure at worst site per mouth for intrabony defects | Measured at Timepoint 1 (from 6 months up to 1 year)
  Secondary outcome
Changes in periodontal probing pocket (PPD) for intrabony defects at site and patient level. | Changes measured from baseline (Timepoint 0) to Timepoint 1( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome
Changes in clinical attachment level (CAL) for intrabony defects at site and patient level. | Changes measured from baseline (Timepoint 0) to Timepoint 1( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome
Changes in horizontal furcation involvement | Changes measured from baseline (Timepoint 0) to Timepoint 1( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome
Changes in vertical CAL for furcation defects | Changes measured from baseline (Timepoint 0) to Timepoint 1( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome
Change in diagnosis of periodontal disease | Changes measured from baseline (Timepoint 0) to Timepoint 1( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome
Radiographic bone levels changes at site level | Changes measured from baseline (Timepoint 0) to Timepoint 1( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome
Radiographic bone levels changes at tooth level | Changes measured from baseline (Timepoint 0) to Timepoint 1( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome
Tooth loss | Changes measured from baseline (Timepoint 0) to Timepoint 1( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome
Correlation of pocket closure to type of surgical approach used (minimally invasive approach, papilla preservation flaps, conventional flaps) | Assessed at Timepoint 1 ( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome- Measured as % of sites with pocket closure (PPD< and = 4mm with no BoP)
Correlation of pocket closure to biomaterials used | Assessed at Timepoint 1 ( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome- Measured as % of sites with pocket closure (PPD< and = 4mm with no BoP)
Correlation of pocket closure to diabetes status | Assessed at Timepoint 1 ( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome- Measured as % of sites with pocket closure (PPD< and = 4mm with no BoP)
Correlation of pocket closure to smoking history | Assessed at Timepoint 1 ( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome- Measured as % of sites with pocket closure (PPD< and = 4mm with no BoP)
Correlation of pocket closure to supportive periodontal therapy frequency | Assessed at Timepoint 1 ( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome- Measured as % of sites with pocket closure (PPD< and = 4mm with no BoP)
Correlation of pocket closure to level of clinician's experience | Assessed at Timepoint 1 ( from 6 months up to 1 year) and Timepoint 2 (through study completion, an average of 2 years)
  Secondary outcome- Measured as % of sites with pocket closure (PPD< and = 4mm with no BoP)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Gkranias, PhD, Principal Investigator — Centre for Oral Clinical Research, QMUL
Locations (1):
- Barts Health NHS Trust Dental Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cortellini P, Buti J, Pini Prato G, Tonetti MS. Periodontal regeneration compared with access flap surgery in human intra-bony defects 20-year follow-up of a randomized clinical trial: tooth retention, periodontitis recurrence and costs. J Clin Periodontol. 2017 Jan;44(1):58-66. doi: 10.1111/jcpe.12638. Epub 2016 Nov 22. PMID 27736011
- [Background] Cortellini P, Tonetti MS. Long-term tooth survival following regenerative treatment of intrabony defects. J Periodontol. 2004 May;75(5):672-8. doi: 10.1902/jop.2004.75.5.672. PMID 15212349
- [Background] Cortellini P, Tonetti MS. Clinical concepts for regenerative therapy in intrabony defects. Periodontol 2000. 2015 Jun;68(1):282-307. doi: 10.1111/prd.12048. PMID 25867990
- [Background] Guerrero A, Griffiths GS, Nibali L, Suvan J, Moles DR, Laurell L, Tonetti MS. Adjunctive benefits of systemic amoxicillin and metronidazole in non-surgical treatment of generalized aggressive periodontitis: a randomized placebo-controlled clinical trial. J Clin Periodontol. 2005 Oct;32(10):1096-107. doi: 10.1111/j.1600-051X.2005.00814.x. PMID 16174275
- [Background] Hamp SE, Nyman S, Lindhe J. Periodontal treatment of multirooted teeth. Results after 5 years. J Clin Periodontol. 1975 Aug;2(3):126-35. doi: 10.1111/j.1600-051x.1975.tb01734.x. PMID 1058213
- [Background] Jepsen S, Topoll H, Rengers H, Heinz B, Teich M, Hoffmann T, Al-Machot E, Meyle J, Jervoe-Storm PM. Clinical outcomes after treatment of intra-bony defects with an EMD/synthetic bone graft or EMD alone: a multicentre randomized-controlled clinical trial. J Clin Periodontol. 2008 May;35(5):420-8. doi: 10.1111/j.1600-051X.2008.01217.x. Epub 2008 Mar 12. PMID 18341601
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of severe periodontitis in 1990-2010: a systematic review and meta-regression. J Dent Res. 2014 Nov;93(11):1045-53. doi: 10.1177/0022034514552491. Epub 2014 Sep 26. PMID 25261053
- [Background] Lang NP, Bartold PM. Periodontal health. J Clin Periodontol. 2018 Jun;45 Suppl 20:S9-S16. doi: 10.1111/jcpe.12936. PMID 29926485
- [Background] Linares A, Cortellini P, Lang NP, Suvan J, Tonetti MS; European Research Group on Periodontology (ErgoPerio). Guided tissue regeneration/deproteinized bovine bone mineral or papilla preservation flaps alone for treatment of intrabony defects. II: radiographic predictors and outcomes. J Clin Periodontol. 2006 May;33(5):351-8. doi: 10.1111/j.1600-051X.2006.00911.x. PMID 16634957
- [Background] Matuliene G, Pjetursson BE, Salvi GE, Schmidlin K, Bragger U, Zwahlen M, Lang NP. Influence of residual pockets on progression of periodontitis and tooth loss: results after 11 years of maintenance. J Clin Periodontol. 2008 Aug;35(8):685-95. doi: 10.1111/j.1600-051X.2008.01245.x. Epub 2008 Jul 23. PMID 18549447